CLINICAL TRIAL: NCT07318116
Title: The Effect of Cabbage Leaf Application on Pain, Physical Function and Quality of Life Levels of Patients With Knee Osteoarthritis
Brief Title: Cabbage Leaf Application in Knee Osteoarthritis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Serap Parlar Kılıç, Prof.Dr, Inonu University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 20/05/2025-592777
Record Dates: First submitted 2025-11-29; First posted 2026-01-05 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Knee Osteoarthritis; Pain
Keywords: Pain; Knee Osteoarthritis; Nursing; Cabbage leaf; Quality of life
MeSH Terms: conditions — Osteoarthritis, Knee; Pain | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The sequence order was generated by computer (Research Randomizer software, version 1.0.0). Unstratified block randomization with varying block sizes will be used to assign patients to three groups. Subsequently, a non-participating staff member will be asked to draw one number from an envelope containing numbers 1 to 90, each representing a patient. The group assignment of the drawn number will determine the patient's group. Using this method, patients will be randomly assigned to the groups. Patients who apply cabbage leaves kept at room temperature, as determined by the literature, will form Experimental Group 1; those who apply traditionally prepared cabbage leaves will form Experimental Group 2; and those who do not receive any cabbage leaf application will form the Control Group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The effect of cabbage leaves on knee pain (Experimental): The sequence order was generated by computer (Research Randomizer software, version 1.0.0). Unstratified block randomization with varying block sizes will be used to assign patients to three groups. Subsequently, a non-participating staff member will be asked to draw one number from an envelope containing numbers 1 to 90, each representing a patient. The group assignment of the drawn number will determine the patient's group. Using this method, patients will be randomly assigned to the groups.
  Patients who apply cabbage leaves kept at room temperature, as determined by the literature, will form Experimental Group 1; those who apply traditionally prepared cabbage leaves will form Experimental Group 2; and those who do not receive any cabbage leaf application will form the Control Group.
  Interventions: Other: Cabbage leaf compress for knee pain

INTERVENTIONS:
Other: Cabbage leaf compress for knee pain — The benefits provided by cabbage leaf compresses have significant potential to enhance individuals' quality of life, facilitate symptom management, and offer an accessible treatment option for a broader patient population. These findings not only support current therapeutic practices but also play a stimulating role in promoting scientific research aimed at developing alternative therapies and holistic health approaches.
  Other Names: Experimental Group 1; Control Group; Experimental Group 2

SUMMARY:
Among non-pharmacological treatment methods, herbal therapies are widely used, and cabbage leaves are recognized for their analgesic and anti-edematous effects. Previous studies indicate that patients often use cabbage leaves for breast engorgement and joint pain, and their strong antioxidant, anticancer, and anti-inflammatory properties have been demonstrated. This study aims to examine the effects of cabbage leaf application on pain, physical function, and quality of life in patients with knee osteoarthritis.

This research is designed as an experimental, mixed-method, randomized controlled trial with a pretest-posttest structure. It will be conducted at the Physical Therapy and Rehabilitation outpatient clinic and inpatient units of Şırnak State Hospital between 01.08.2025 and 01.08.2026. A total of 90 patients will be included and randomly assigned to three groups of 30 participants: those receiving room-temperature cabbage leaf application (Experimental Group 1), those receiving traditionally prepared cabbage leaf application (Experimental Group 2), and those receiving no cabbage leaf application (Control Group).

Data will be collected using the Patient Information Form, A-VAS, WOMAC, and the Mini-OAKHQoL-TR Scale. Experimental groups will receive a daily 2-hour cabbage leaf application for 4 weeks, while the control group will receive routine care only. Measurements will be conducted at weeks 1 and 4.

Data will be analyzed using SPSS 22.0. Descriptive statistics will summarize the sample. Normality will be tested with the Kolmogorov-Smirnov test. For normally distributed data, independent t-test, paired t-test, ANOVA, and ANCOVA will be used; for non-normal data, Mann-Whitney U, Kruskal-Wallis H, Wilcoxon signed-rank, and Friedman tests will be applied.

This study aims to contribute evidence supporting non-pharmacological interventions as alternative or complementary approaches in managing joint and knee pain. Such applications may help reduce healthcare costs, decrease hospitalization rates, improve accessibility, save time, and provide an economical therapeutic option within clinical practice.

DETAILED DESCRIPTION:
Osteoarthritis, which develops under the influence of genetic, mechanical, or biochemical factors, is a chronic inflammatory degenerative joint disease characterized by morphological alterations of the synovial membrane and joint capsule, including synovial inflammation, progressive cartilage degradation, the formation of osteophytes, and subchondral bone sclerosis, particularly in weight-bearing joints. Due to the greater degree of degeneration in weight-bearing joints, the knee is the most commonly affected joint in symptomatic osteoarthritis. In addition to the knee, the hip, spine, hand, foot, and fingers are among the other joints frequently involved. Progressive cartilage loss in the knee joint leads to limitations in range of motion, severe chronic pain, and significant muscle atrophy. Knee pain-often sharp, dull, continuous, or intermittent-is one of the most common symptoms associated with osteoarthritis. Crepitus during physical examination, stiffness and swelling, restricted motion, morning stiffness, and muscle weakness are also frequently observed. Pain that initially occurs during activity may progress to pain at rest as the disease advances, making it one of the leading reasons for clinical visits.

According to 2019 data, approximately 528 million individuals worldwide were living with osteoarthritis, representing a 113% increase since 1990. Nearly 73% of patients with osteoarthritis are over 55 years of age, and approximately 60% are women. As osteoarthritis is more common among older adults (with about 70% of cases occurring in individuals over 55 years of age), global prevalence is expected to rise with population aging. Based on data from the Turkish Statistical Institute (TUIK), 11.2% of the population in Türkiye reported arthritis-related problems in 2019.

Several risk factors contributing to the development and progression of OA have been identified. The onset and progression of the disease are influenced by genetics, age, sex, nutrition, obesity, bone density, joint stress resulting from sports activities, smoking, ethnicity, physical inactivity, occupational joint strain, and trauma. Moreover, more than 25% of osteoarthritis cases are accompanied by comorbid conditions such as obesity, diabetes, pulmonary and cardiovascular diseases, hypertension, metabolic and musculoskeletal disorders, and depression. The chronic pain and stiffness experienced by individuals with osteoarthritis lead to physical limitations that impair daily living activities, result in inadequate self-care, deteriorate functional status, disrupt social relationships, and ultimately contribute to decreased quality of life. Age-related increases in musculoskeletal conditions within society negatively affect functional capacity, quality of life, and healthcare costs. Education, weight management, and regular exercise are effective strategies for improving quality of life. Challenges in nutrition, transportation, elimination, and social interaction further impair quality of life among older individuals. Therefore, improving quality of life should be prioritized in the self-management of osteoarthritis.

Although there is no direct cure for osteoarthritis, treatment strategies aim to reduce symptoms, slow disease progression, minimize the negative impact on mobility and quality of life, and lessen healthcare needs. Pharmacological treatments include analgesics, anti-inflammatory agents, and opioids, while surgical interventions involve arthroscopy, osteotomy, and total knee replacement. Non-pharmacological therapies constitute one of the strongly recommended components in osteoarthritis management, particularly in knee osteoarthritis, as emphasized by the European Society for Clinical and Economic Aspects of Osteoporosis, Osteoarthritis and Musculoskeletal Diseases (ESCEO). Strongly recommended approaches include patient education, weight loss when applicable, and structured exercise programs consisting of aerobic and strengthening exercises, alongside lifestyle modifications. Additionally, modalities suggested by the European League Against Rheumatism (EULAR)-such as laser therapy, spa therapy, pulsed electromagnetic field therapy, acupuncture, transcutaneous electrical nerve stimulation (TENS), herbal remedies, and vitamin supplementation-are commonly used non-pharmacological treatment options.

Herbal remedies are widely recommended as complementary and supportive treatments in many healthcare systems across the world. Some self-care guidelines frequently advise the use of bandages or compresses for osteoarthritis symptoms. Among these traditional practices, cabbage leaf compresses have been used for centuries. Leaves from white or Savoy cabbage are applied to the painful knee joint for several hours to reduce pain. The health-promoting properties of cabbage leaves have long been recognized, and they have been used to treat various conditions, including breast engorgement. Cabbage leaves are rich in dietary fiber, vitamin C, vitamin K, folate, manganese, iodine, potassium, beta-carotene, and calcium. They are also known to possess strong antioxidant, anticancer, and anti-inflammatory properties. The sulfur compounds in cabbage leaves are believed to help alleviate pain and swelling. Their analgesic effects are attributed to physiological mechanisms such as dilation of capillaries, reduction of tissue congestion, decreased edema, localized anesthetic effects, and reduction in muscle spasticity and stiffness.

A quasi-experimental pretest-posttest study involving 60 elderly patients aged 60-85 with joint pain demonstrated that cabbage leaf compresses effectively reduced pain levels, as indicated by a decrease from a pretest mean of 7.60 to a posttest mean of 2.17. Another single-group pretest-posttest study evaluating the effectiveness of cabbage compresses over three weeks in 50 older adults found a significant decrease in mean pain scores from 3.58±0.70 to 0.18±0.38 (p < 0.001). Similarly, a randomized controlled trial in patients with knee OA revealed significant reductions in pain, improvements in functional limitations after four weeks, and enhancements in overall quality of life at twelve weeks following cabbage leaf treatment. Another randomized study involving 60 patients with moderate to severe OA (Kellgren-Lawrence grade 3-4) and moderate Oxford Knee Scores assigned participants to three intervention groups: cooling gel pack (20 minutes daily), diclofenac gel applied four times daily as a control, and cabbage leaf application for 1 hour daily. All participants recorded their pain using the Numerical Rating Scale (NRS) and their Oxford Knee Scores, with evaluations conducted weekly and after four weeks. The findings demonstrated that cabbage leaf application and cooling gel packs yielded comparable improvements in NRS and Oxford Knee Scores, both outperforming diclofenac gel.

Additionally, cabbage leaves have been shown to effectively reduce breast engorgement and associated pain and discomfort. Despite their common use, the literature indicates that research on cabbage leaf compresses in patients with knee osteoarthritis remains limited. Barriers such as restricted access to healthcare facilities, economic challenges, cultural variations, and differences in the application of herbal treatments contribute to this gap. This study aims to contribute to healthcare practice by supporting the incorporation of cabbage-a low-cost, widely accessible, and easy-to-use plant-into non-pharmacological treatment options for patients.

Evidence from the relevant literature indicates that cabbage leaf compresses reduce pain and swelling, and improve quality of life in patients experiencing joint pain, knee osteoarthritis, and breast engorgement. Integrating alternative treatment approaches-such as Traditional and Complementary Medicine-into clinical practice alongside pharmacological therapy may provide valuable insights into the role of herbal medicine in pain management. Supporting the incorporation of cabbage leaf applications into holistic treatment plans for conditions such as joint and knee pain or breast engorgement offers patients an economical, easily applicable, accessible, comfortable, single-use, and non-pharmacological option, particularly in resource-limited settings.

Cabbage leaf application may contribute to scientific knowledge by providing evidence of its natural analgesic properties, promoting alternative pain management strategies, and encouraging further research into plant-based therapeutic agents for pain relief. Educating healthcare professionals on cabbage leaf application may also enable them to recommend such evidence-based, beneficial practices to patients. Furthermore, identifying the physical or chemical effects of cabbage on pain and other symptoms could facilitate the development of new products or materials within future research projects.

Based on the anticipated outcomes of the planned study, cabbage leaf application may serve as an alternative treatment method that improves patient symptoms and quality of life by offering an economical, easy-to-apply, and effective approach to acute pain management. From a healthcare perspective, it may also help reduce treatment costs and decrease the time patients spend in hospital settings. In addition, depending on the study results, future research may extend beyond physical therapy and obstetrics clinics to explore its applicability in other populations-particularly oncology and palliative care patients-by examining its potential effects on symptoms that arise in these clinical contexts.

ELIGIBILITY:
Inclusion Criteria:

* Experiencing knee pain due to osteoarthritis for at least 6 months
* Diagnosed with knee osteoarthritis by a physician according to the American College of Rheumatology (ACR) criteria
* Having a pain score of 4 or higher on the Visual Analog Scale (VAS)
* Aged 18 years or older
* No allergy to cabbage or other herbal products
* Able to speak Turkish and having no communication difficulties
* Volunteering to participate in the study

Exclusion Criteria:

* Those with poor mental status
* Those using pain-relieving medication during the cabbage leaf application period
* Those with a history of surgical operation on the application area (knee region) within the past year
* Those with infection, wounds, cellulitis, or skin disease in the application area
* Those with any peripheral vascular disease in the application area
* Those who have experienced significant knee trauma within the past six months
* Those who have received intra-articular steroid injections within the past six months
* Those with inflammatory joint disease
* Those who developed knee osteoarthritis due to injury or infection
* Those with pain related to secondary arthritis (e.g., post-traumatic or inflammatory arthritis)
* Those with asthma, liver, or kidney disease
* Pregnant or breastfeeding women
* Those with psychological or physical disorders
* Those with physical disabilities in the lower extremities
* Patients who do not agree to participate in the study will not be included in the sample.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2026-01-10 (Actual); Study Completion 2026-02-25 (Estimated)

PRIMARY OUTCOMES:
Change in Knee Pain Severity | 1 month
  Description: Knee pain severity will be measured using the Visual Analog Scale/VAS (0-10). Change in VAS pain score from baseline to Week 4 will be assessed.
  Unit of Measure: Points on a 0-10 scale
Change in Physical Function | 1 month
  Description: Physical function will be assessed using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Physical Function Subscale. Change from baseline to Week 4 will be evaluated.
  Unit of Measure: Points on WOMAC scale (0-96)
Change in Quality of Life | 1 month
  Description: Quality of Life in Lower Extremity Osteoarthritis (MiniOAKHQoL-TR) questionnaire will be used for measurement. Change from baseline to week 4 will be evaluated.
  Unit of Measure: Quality of Life in Lower Extremity Osteoarthritis (MiniOAKHQoL-TR) scores (0-200)

CONTACTS AND LOCATIONS:
Overall Officials: Feyzi DOĞRU, Ass. Prof, Principal Investigator — Malatya Turgut Özal University / Faculty of Medicine / Department of Basic Medical Sciences / Division of Physiology; Serap PARLAR KILIÇ, Prof. Dr., Study Director — Inonu Unıversty; Mehmet Hayrullah ÖZTÜRK, Phd Student, Study Chair — Sırnak Unıversty
Locations (1):
- Şirnak State Hospital, Şirnak, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This information can be shared upon reasonable request after the study is completed.

REFERENCES:
- [Result] Chobpenthai T, Arunwatthanangkul P, Mahikul W. Efficacy of Cabbage Leaf versus Cooling Gel Pad or Diclofenac Gel for Patients with Knee Osteoarthritis: A Randomized Open-Labeled Controlled Clinical Trial. Pain Res Manag. 2022 Jun 8;2022:3122153. doi: 10.1155/2022/3122153. eCollection 2022. PMID 35719197
- [Result] Ozkaya M, Korukcu O. Effect of cold cabbage leaf application on breast engorgement and pain in the postpartum period: A systematic review and meta-analysis. Health Care Women Int. 2023 Mar;44(3):328-344. doi: 10.1080/07399332.2022.2090567. Epub 2022 Jun 29. PMID 35766462
- [Result] Lauche R, Graf N, Cramer H, Al-Abtah J, Dobos G, Saha FJ. Efficacy of Cabbage Leaf Wraps in the Treatment of Symptomatic Osteoarthritis of the Knee: A Randomized Controlled Trial. Clin J Pain. 2016 Nov;32(11):961-971. doi: 10.1097/AJP.0000000000000352. PMID 26889617